CLINICAL TRIAL: NCT00224029
Title: A Multi-center, Open-label, Dose-titration Pilot Study Evaluating the Efficacy and Safety of Oxybutynin Transdermal Systems in Patients With Neurogenic Bladder Resulting From Spinal Cord Injury
Brief Title: A Study Evaluating Oxybutynin in Patients With Neurogenic Overactive Bladder Associated With a Neurological Condition
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Watson Pharmaceuticals (Industry)
Responsible Party: Gary Hoel, RPh, PhD, Watson Laboratories, Inc
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OXY0401
Record Dates: First submitted 2005-09-13; First posted 2005-09-22 (Estimated); Results first posted 2010-04-30 (Estimated); Last update posted 2010-04-30 (Estimated); Status verified 2010-04

CONDITIONS: Detrusor Hyperreflexia
MeSH Terms: interventions — oxybutynin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Oxybutynin transdermal system (Experimental): Oxybutynin transdermal system 3.9 mg/day, 7.8 mg/day, 9.1 mg/day or 11.7 mg/day dosing
  Interventions: Drug: Oxybutynin transdermal system

INTERVENTIONS:
Drug: Oxybutynin transdermal system — 3.9 mg/day, 7.8 mg/day, 9.1 mg/day or 11.7 mg/day transdermal per titration
  Other Names: Oxytrol

SUMMARY:
This study will evaluate the efficacy and safety of an anticholinergic drug treatment administered by transdermal patch to treat overactive bladder in adults who have spinal cord injury.

DETAILED DESCRIPTION:
The Dose Titration Period began with a 3.9 mg/day or 7.8 mg/day as a starting dose after the completion of a 3-day diary for baseline evaluations, including urodynamic testing. The clean intermittent catheterization (CIC) frequency remained constant throughout the Dose Titration Period. The dose was adjusted every two weeks during the Dose Titration Period by increasing one dose level, at the investigator's discretion, based on the patient's symptoms. If a patient achieved complete continence and reported tolerable or absence of side effects, the patient was continued at that dose for the duration of the 8-week Titration Period. If a patient reported unacceptable side effects, the dose was reduced by one level. This reduced dose was considered the maximum tolerable dose for the patient and the patient continued at that dose for the duration of the 8-week Titration Period. The dose levels evaluated were 3.9 mg/day, 7.8 mg/day, 9.1 mg/day, and 11.7 mg/day. Of the 22 subjects in the modified intent-to-treat population evaluated for efficacy, 0 were in the 3.9 mg/day dose group, 3 were in the 7.8 mg/day dose group, 8 were in the 9.1 mg/day dose group, and 11 were in the 11.7 mg/day dose group.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age at day of consent;
* Is a male, or is a non-pregnant non-lactating female who is either of non-child-bearing potential, or is using adequate means of birth control;
* Has a h/o of urinary incontinence from neurogenic bladder of spinal cord injury etiology;
* Has impairment based on the American Spinal Injury Association (ASIA);
* Use clean intermittent catheterization;
* Has urinary incontinence between scheduled catheterization;
* Capable of understanding and complying with the protocol.

Exclusion Criteria:

* Have one or more treatable conditions, other than neurogenic bladder dysfunction, that may cause urinary incontinence or urgency;
* Have any medical condition that precludes their participation in the study, or may confound the outcome of the study;
* History of major lower urinary tract surgery, procedures;
* Has an active skin disorder, affecting TDS application site areas;
* Hypersensitivity to the investigational drug;
* Has participated in any study involving administration of an investigational compound within 30 days before this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2004-12; Primary Completion 2005-12 (Actual); Study Completion 2008-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gary Hoel, RPh, PhD, Study Director — Watson Laboratories, Inc.
Locations (6):
- United States (6):
  - Atlanta, Georgia
  - The Bronx, New York
  - Chapel Hill, North Carolina
  - Charlotte, North Carolina
  - Dallas, Texas
  - Houston, Texas

REFERENCES:
- [Result] Kennelly MJ, Lemack GE, Foote JE, Trop CS. Efficacy and safety of oxybutynin transdermal system in spinal cord injury patients with neurogenic detrusor overactivity and incontinence: an open-label, dose-titration study. Urology. 2009 Oct;74(4):741-5. doi: 10.1016/j.urology.2009.05.008. Epub 2009 Jul 22. PMID 19628264

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: washout of previous anticholinergic therapy during the screening period
Period: Overall Study
Arm/Group | Oxybutynin Transdermal System
Started | 24
Completed | 18
Not Completed | 6
Not completed — Lost to Follow-up | 1
Not completed — Withdrawal by Subject | 4
Not completed — Other | 1

BASELINE CHARACTERISTICS:
Arm/Group | Oxybutynin Transdermal System
Number analyzed (Participants) | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 24
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 41.9 (10.35)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 21
Region of Enrollment [Number; unit: participants]
  United States | 24

OUTCOME MEASURES:

1. Primary Outcome: Average Number of Catheterizations Without Leaking Per Day
Description: Baseline in number of daily catheterizations without leaking per day as recorded in a 3-day urinary diary.
Time Frame: 8 weeks
Population: The number of participants for analysis is determined by Last Observation Carried Forward (LOCF.
Measure: Mean (Standard Deviation); unit: Number of Dry Catheterizations per Day
Arm/Group | Oxybutynin Transdermal System
Number analyzed (Participants) | 22
Number of Dry Catheterizations per Day
  Baseline at Week 0 | 2.4 (1.8)
  Change from baseline at Week 8 | 1.5 (2.2)

2. Secondary Outcome: Patch Adhesion
Time Frame: 8 weeks
Reporting Status: Not Posted

3. Secondary Outcome: Urodynamic Measurements
Time Frame: 8 weeks
Reporting Status: Not Posted

4. Secondary Outcome: Urinary Leakage and Catheterization Data
Time Frame: 8 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 8 weeks
Arm/Group | Oxybutynin Transdermal System
Serious Adverse Events (participants affected / at risk) | 0/24
Other Adverse Events (participants affected / at risk) | 11/24
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oxybutynin Transdermal System (N=24)
Dry mouth (Gastrointestinal disorders) | 2 (5)
Headache (General disorders) | 2 (2)
Infection urinary tract (Renal and urinary disorders) | 3 (3)
Sweat (Skin and subcutaneous tissue disorders) | 2 (3)
Vision abnormal (Eye disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less